CLINICAL TRIAL: NCT02915887
Title: The Short-term Effect of Cervical Taping on Neck Pain, Disability and Kinematics in Patients With Chronic Neck Pain: A Non-randomised Clinical Trial
Brief Title: The Effect of Cervical Taping on Neck Pain and Kinematics in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Hilla Sarig Bahat, Dr, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HillaUHaifa
Record Dates: First submitted 2016-09-18; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Neck Pain; Cervical Pain; Chronic Pain
Keywords: neck pain; chronic; taping; kinematics; motion analysis; physiotherapy
MeSH Terms: conditions — Neck Pain; Chronic Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cervical taping (Experimental): Participants received treatment including elastic taping application to the neck. They were assessed 3 times: Pre taping, 20 minutes post-taping on day 1, and 7 days post-taping.
  Interventions: Other: Cervical Taping

INTERVENTIONS:
Other: Cervical Taping — Kinesio®Tex Tape 23 was used in this study. Two strips of tape were applied. The first layer was a Y-shaped strip with 2 tails on 2 sides of the cervical vertebrae, placed over the posterior cervical extensor muscles and applied from the insertion to origin. The second strip was an I-shaped approximately 20cm long, transversally applied over the C5-C7 vertebra with a tension-on-base technique in a space correction technique.

SUMMARY:
Objective: This study examined the effects of elastic tape applied to the neck on patients experiencing chronic neck pain.

Background: Neck pain is often persistent or recurrent. Various treatments have been described, including exercises and manual therapy. Taping is commonly used clinically in the management of neck pain, however research in this field is sparse.

Methods: Elastic tape was applied over the posterior cervical extensor muscles from insertion to origin on patients experiencing chronic neck pain. Patients were assessed pre-taping, immediately post-taping, and one week post-taping and did not receive additional physiotherapy during the study.

Subjective measures included the Visual Analogue Scale (VAS) for pain intensity, the Neck Disability Index (NDI) to determine the level of disability in daily living, and the Tampa Scale of Kinesiophobia (TSK) to assess fear of movement or re-injury. Objective outcome measures included cervical range of motion, velocity, smoothness, and accuracy of cervical motion. These kinematic measures were collected using a customised virtual reality system designed to evaluate neck motion disorders.

DETAILED DESCRIPTION:
Neck pain is a common disorder, affecting 30-50% of the general population annually, comprising approximately 25% of the patients receiving physiotherapy in outpatient clinics. Symptoms include pain and stiffness in the neck, headache, dizziness, and pain radiating to the shoulders or upper limbs. Physical impairments associated with neck pain can include decreased cervical range of motion (ROM), increased fatigability, compromised strength and endurance of the cervical muscles, and impaired sensorimotor control.

A variety of Physiotherapeutic interventions have been described for the treatment of neck pain. Taping is a passive technique, widely used for the treatment of sport injuries, muscle imbalance, and impaired neural control. Clinically, taping is used for neck pain in spite of lack of research regarding its effectiveness. In addition, the mechanism by which elastic tape application affects tissue and function is yet unknown, but various effects have been described such as the ability to increase ROM, facilitate muscles and proprioception, and decrease pain.

A literature search retrieved only 3 relevant studies examining the use and efficacy of elastic tape on the cervical spine. Gonzalez-Iglesias et al. (2009) conducted a randomized trial in whiplash patients, Karatas et al. (2012) studied the effect of taping in surgeons with cervical pain after performing surgery, and Saavedra-Hernandez et al (2012)- in patients with mechanical neck pain.

All three studies demonstrated short-term effectiveness of elastic taping on pain relief and cervical ROM. However, all samples were small, of mostly young participants, and effect size was not described. Reported changes were small implying that further research is needed.

The objective of this study was to evaluate the short-term effect of cervical elastic taping on pain intensity, disability and neck kinematics in patients with chronic neck pain.

Materials and Methods

This study was a non-controlled trial with a pre-post test design and a single intervention group. Ethics approval was obtained from the ethics committee, the Faculty of Social welfare and Health Sciences at the University of Haifa, and from the Helsinki committee at Rambam Health Care Campus Helsinki Committee.

Participants

A convenience sample of 27 individuals, 13 males and 14 females, was recruited via electronic media. Inclusion criteria were (a) chronic neck pain (>3 months), with or without referral to the upper limb; (b) age of 18 years or more; (c) pain intensity≥ 30% on Visual Analogue Scale (VAS). Subjects were excluded if they had physiotherapy in the previous 2 months, known skin allergy to the tape, evidence for active vestibular disorders, medical conditions that may affect performance such as Rheumatic Arthritis, Diabetes Mellitus, neurological disorders, head injuries, lower limb pathologies, local or systemic infections, inability to communicate and provide informed consent, unstable fracture/dislocation, post-orthopaedic surgery in the upper body or spine, and pregnancy. Following screening, each participant signed a consent form.

Virtual Reality Assessment

A neck virtual reality (VR) system was used to assess cervical motion kinematics by the protocol of Sarig-Bahat et al. (2010). This system included off-the-shelf hardware and customized software. Hardware included a head-mounted display with a built-in tracker. Virtual environment software was developed using Unity-pro software, version 3.40f520.

Cervical motion was elicited by interaction with images during a video game displayed on the two monitors embedded in the HMD. All dynamic motion data was recorded during the VR session and analysed by the software in real-time. During the game, the participant acts as a pilot flying an airplane. The position of the airplane was controlled by the participant's head motion. Yellow targets were displayed on the HMD monitors and the participant had to contact them within 5 seconds by aligning the airplane with the virtual target. Once the target was contacted, a new target would appear at a random location and the player's task was to move towards it. Based on this principle, the VR assessment included (a) evaluating cervical ROM, (b) cervical motion velocity, and (c) cervical motion accuracy during a smooth head pursuit task.

Taping Technique

Kinesio®Tex Tape 23 was used in this study. Two strips of tape were applied: The first layer was a Y-shaped strip with 2 tails on 2 sides of the cervical vertebrae, placed over the posterior cervical extensor muscles and applied from the insertion to origin. The second strip was an I-shaped approximately 20cm long, transversally applied over the C5-C7 vertebra with a tension-on-base technique in a space correction technique.

Study Procedure

Patients were screened by inclusion and exclusion criteria. The physiotherapist performing the assessments and taping techniques was a qualified physiotherapist with 13 years of clinical experience in musculoskeletal physiotherapy and was a qualified Kinesio® taping practitioner.

Each patient was assessed 3 times: pre- and 20 minutes post-taping on day 1, and in a follow-up assessment 7 days later.

Following the subjective examination and completion of the questionnaires, an explanatory VR session was provided to minimize training effects and to reach a stable level of VR control. Patients were evaluated in upright sitting position, with the trunk strapped to the back of a rigid chair to eliminate thoracic motion. Calibration was performed at each session for each participant, as instructed by the manufacturer. Each VR evaluation took up to 15 minutes. Breaks were provided when needed. Following the assessment, tape was applied. After a washout period 20 minutes post-taping application, the second examination was performed. No other physiotherapy procedures were provided. Patients were instructed to maintain the elastic tape for up to 5 days. They were instructed to remove the tape if symptoms were aggravated or if any topical irritation appeared. The third examination was one-week after the initial examination and included VR assessment without tape application.

A paired-samples t-test was used to evaluate the pre-post differences in studied outcome measures. Two paired-sample t-tests were run: pre- vs. immediate post-, and pre- vs. one week post-taping. Significance level was set at 5%. Cohen's d was calculated to determine the effect size. Data were analyzed using the SPSS software, version 17.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (>3 months), with or without referral to the upper limb;
* Age of 18 years or more;
* Pain intensity ≥ 30% on Visual Analogue Scale (VAS).

Exclusion Criteria:

* Subjects were excluded if they had physiotherapy in the previous 2 months, known skin allergy to the tape, evidence for active vestibular disorders, medical conditions that may affect performance such as Rheumatic Arthritis, Diabetes Mellitus, neurological disorders, head injuries, lower limb pathologies, local or systemic infections, inability to communicate and provide informed consent, unstable fracture/dislocation, post-orthopaedic surgery in the upper body or spine, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity was measured by theVisual Analogue Scale (VAS, 0-100mm) | One week
  The Visual Analogue Scale (VAS) was used to measure neck pain intensity (0- 100mm).
Cervical range of motion was measured by the neck VR system (ROM, degrees) | One week
  Cervical range of motion was measured to four directions- flexion, extension, right and left rotation, during the VR assessment.

SECONDARY OUTCOMES:
Cervical motion accuracy was measured by the VR system (Accuracy, degrees). | one week
  Cervical motion accuracy was collected in the VR accuracy module. It was defined as the difference in degrees between target and player position at each given sample to provide values for accumulated accuracy error in degrees.
Self-reported disability was measured using the Neck Disability Index (NDI, 0-100%) | One week
  Disability due to neck pain was measured using the neck disability index (NDI)
Fear of movement was assessed using the TAMPA Scale of Kinesiophobia (TSK, 0-68) | One week
  Tampa Scale of Kinesiophobia (TSK) was used to assess fear of movement or re-injury. TSK was found to be associated with measures of behavioral avoidance and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Sarig Bahat, PT, PhD, Principal Investigator — Department of Physical Therapy, University of Haifa
Locations (1):
- The Faculty of Social Welfare and Health Sciences, Haifa, Haifa District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald, Taping techniques principles and practice. second edition ed. 2004: Elsevier limited.
- [Background] Gonzalez-Iglesias J, Fernandez-de-Las-Penas C, Cleland JA, Huijbregts P, Del Rosario Gutierrez-Vega M. Short-term effects of cervical kinesio taping on pain and cervical range of motion in patients with acute whiplash injury: a randomized clinical trial. J Orthop Sports Phys Ther. 2009 Jul;39(7):515-21. doi: 10.2519/jospt.2009.3072. PMID 19574662
- [Background] Kalichman L, Vered E, Volchek L. Relieving symptoms of meralgia paresthetica using Kinesio taping: a pilot study. Arch Phys Med Rehabil. 2010 Jul;91(7):1137-9. doi: 10.1016/j.apmr.2010.03.013. PMID 20537313
- [Background] Karatas N, Bicici S, Baltaci G, Caner H. The effect of Kinesiotape application on functional performance in surgeons who have musculo-skeletal pain after performing surgery. Turk Neurosurg. 2012;22(1):83-9. doi: 10.5137/1019-5149.JTN.5377-11.1. PMID 22274976
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Background] Halseth T, McChesney JW, Debeliso M, Vaughn R, Lien J. The effects of kinesio taping on proprioception at the ankle. J Sports Sci Med. 2004 Mar 1;3(1):1-7. eCollection 2004 Mar. PMID 24497814
- [Background] Saavedra-Hernandez M, Castro-Sanchez AM, Arroyo-Morales M, Cleland JA, Lara-Palomo IC, Fernandez-de-Las-Penas C. Short-term effects of kinesio taping versus cervical thrust manipulation in patients with mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2012 Aug;42(8):724-30. doi: 10.2519/jospt.2012.4086. Epub 2012 Apr 20. PMID 22523090
- [Background] Sarig Bahat H, Weiss PL, Laufer Y. The effect of neck pain on cervical kinematics, as assessed in a virtual environment. Arch Phys Med Rehabil. 2010 Dec;91(12):1884-90. doi: 10.1016/j.apmr.2010.09.007. PMID 21112430